CLINICAL TRIAL: NCT00038753
Title: Vision In Preschoolers Study (VIP Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Eye Institute (NEI) (NIH)
Purpose: Diagnostic
Other Study IDs: NEI-85
Record Dates: First submitted 2002-06-04; First posted 2002-06-05 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Amblyopia; Strabismus; Refractive Error
Keywords: vision screening
MeSH Terms: conditions — Amblyopia; Strabismus; Refractive Errors | interventions — Vision Screening

INTERVENTIONS:
Procedure: Vision Screening

SUMMARY:
To identify vision-screening tests that can accurately predict those three- and four-year old preschoolers who would benefit from a comprehensive vision examination because of signs of amblyopia, strabismus, and/or significant refractive error.

DETAILED DESCRIPTION:
The Vision In Preschoolers (VIP) Study is a multi-center, multidisciplinary, prospective clinical study to evaluate screening tests for identifying preschool children in need of comprehensive eye examinations. The primary goal of the VIP Study is to identify an effective and efficient battery of screening tests that has high sensitivity and specificity in identifying preschoolers in need of further evaluation for amblyopia, strabismus and/or significant refractive error.

The VIP Study is designed in three-phases.

Phase I activities will establish which screening tests perform well when administered by licensed eye care professionals (pediatric optometrists and pediatric ophthalmologists) in a population of 1000 Head Start preschoolers at high risk for the targeted vision disorders.

Phase II activities will provide evaluation of the tests' performance when administered by pediatric nurses and lay people on a high risk population of 1000 Head Start preschoolers. Each child will be tested twice with each screening test - once by a pediatric nurse and once by a lay screener. Tests selected for Phase II will be determined by the outcome of Phase I.

Phase III activities will evaluate the performance of the tests in identifying individuals with specific vision disorders in a general population of (6400) Head Start preschoolers. The category of screening personnel and the specific screening tests used in Phase III will be determined by the outcome of Phases I and II.

ELIGIBILITY:
Children enrolled in Head Start who are between the ages of 3 years 0 months and 4 years 11 months of age.

Ages: 36 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - University of California, Berkeley School of Optometry, Berkeley, California
  - New England College of Optometry, Boston, Massachusetts
  - The Ohio State University College of Optometry, Columbus, Ohio
  - Oklahoma Northeastern State University College of Optometry, Tahlequah, Oklahoma
  - Pennsylvania College of Optometry, Philadelphia, Pennsylvania